CLINICAL TRIAL: NCT06646354
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group, Phase 3 Trial to Evaluate the Efficacy and Safety of Co-administrated HODO-2224-1 and HODO-2224-2 in Patients With Essential Hypertension and Primary Hypercholesterolemia
Brief Title: To Evaluate the Efficacy and Safety of Co-administrated HODO-2224-1 and HODO-2224-2 in Patients With Essential Hypertension and Primary Hypercholesterolemia
Acronym: HODO-2224
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD_CARE_002
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Primary Hypercholesterolaemia
MeSH Terms: conditions — Hypertension | interventions — Ezetimibe; candesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HODO-2224-1+HODO-2224-2+HODO-2224-4 (Experimental): Oral tablet, QD
  Interventions: Drug: Ezetimibe/Rosuvastatin/Candesartan/Amlodipine
- HODO-2224-1+HODO-2224-4+HODO-2224-5 (Active Comparator): Oral tablet, QD
  Interventions: Drug: Candesartan/Amlodipine
- HODO-2224-2+HODO-2224-3+HODO-2224-6 (Active Comparator): Oral tablet, QD
  Interventions: Drug: Candesartan/Rosuvastatin/Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe/Rosuvastatin/Candesartan/Amlodipine — PO, QD, 8 weeks
  Arms: HODO-2224-1+HODO-2224-2+HODO-2224-4
Drug: Candesartan/Amlodipine — PO, QD, 8 weeks
  Arms: HODO-2224-1+HODO-2224-4+HODO-2224-5
Drug: Candesartan/Rosuvastatin/Ezetimibe — PO, QD, 8 weeks
  Arms: HODO-2224-2+HODO-2224-3+HODO-2224-6

SUMMARY:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel group, Phase 3 trial to Evaluate the Efficacy and Safety of Co-administrated HODO-2224-1 and HODO-2224-2 in Patients with Essential Hypertension and Primary Hypercholesterolemia

DETAILED DESCRIPTION:
This trial is a phase 3 study to evaluate the efficacy and safety of Co-administrated HODO-2224-1 and HODO-2224-2 in Patients with Essential Hypertension and Primary Hypercholesterolemia.

This is multi-center, double-blind, Active-controlled, parallel-group, phase 3 study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19
* Patients with Essential Hypertension and Primary Hypercholesterolemia

Exclusion Criteria:

* Patients with differences between arms greater than 20 mmHg for mean sitSBP or 10 mmHg for mean sitDBP
* Patients with mean sitSBP ≥ 180 mmHg or mean sitDBP ≥ 110 mmHg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | baseline and week 8
  LDL-C change at Week 8 compared HODO-2224-1 + HODO-2224-4 + HODO-2224-5 with HODO-2224
Mean sitting systolic blood pressure (MSSBP) | baseline and week 8
  MSSBP change at week 8 compared HODO-2224-2 + HODO-2224-3 + HODO-2224-6 with HODO-2224

SECONDARY OUTCOMES:
change of other Lipid profile | 0, 4, 8 weeks
  change of other Lipid profile

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No